CLINICAL TRIAL: NCT05160376
Title: Efficacy of Guided and Unguided Online Self-help Psychological Intervention for Improving Depressive and Anxiety Symptoms: A Pilot Randomized Controlled Trial
Brief Title: Efficacy of Guided and Unguided Online Self-help Psychological Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY018
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Online Self-help Transdiagnostic Psychological Intervention; Anxiety; Depression
Keywords: Online Self-help; Online Psychological Intervention; Unguided Online Self-help; Guided Online Self-help; Transdiagnostic intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Intervention Group (Experimental): The participants in the guided intervention group will receive feedback calls (approximately 15 minutes) on participants' progress from a clinical psychology trainee or an undergraduate trained psychology student under the supervision of a clinical psychology professor, after each online self-help intervention session. The participants in the guided intervention group will also receive an email reminder and text message if the participants have not completed the required session of that week on the 5th, 6th, and 7th of the same week. Technical supports are available.
  Interventions: Other: Self-help CBT with email reminder and text message; Other: Feedback calls on participants' progress
- Unguided Intervention Group (Experimental): The participants in the unguided intervention group will not receive the aforementioned feedback calls. The participants in the unguided intervention group will only receive an email reminder and text message if the participants have not completed the required session of that week on the 5th, 6th, and 7th of the same week. Technical supports are available.
  Interventions: Other: Self-help CBT with email reminder and text message
- Wait-list Control Group (No Intervention): The waitlist control group will not receive any online self-help intervention. Unguided intervention will be provided to the waitlist control group after both the Post-treatment Assessment Phrase are finished.

INTERVENTIONS:
Other: Self-help CBT with email reminder and text message — An online transdiagnostic self-help intervention that is delivered through an online mental health platform.
  Email reminder and text message will be sent to remind participant to complete the module
  Arms: Guided Intervention Group; Unguided Intervention Group
Other: Feedback calls on participants' progress — Feedback calls (approximately 15 minutes) on participants' progress from a clinical psychology trainee or an undergraduate trained psychology student under the supervision of a clinical psychology professor
  Arms: Guided Intervention Group

SUMMARY:
This study will examine the efficacy of guided and unguided online transdiagnostic self-help cognitive behavioral therapy (CBT) for reducing anxiety and/or depression symptoms in Hong-kong residents. Numerous literature demonstrates online self-help interventions' efficacy on depression and anxiety. Nonetheless, existing research overlooks the mechanism of change, the online treatment outcome's potential predictors, and the effect of therapist's guidance on participants' treatment expectancy and its mediating effect on treatment outcome, which are essential to optimize intervention's efficacy.

96 Hong-kong residents, aged 18-65, with mild to moderate anxiety and/or depression will be recruited. Eligible participants will be randomly assigned to either guided group (Group-1) or unguided group (Group-2) or waitlist control group (Group-3) in a 1:1:1 ratio. Group-1 will receive weekly manualized progress feedback from trained researchers under supervision, after each weekly treatment. Group-2 will not receive the aforementioned feedback. Group-1 and Group-2 will receive reminders on the 5th, 6th and 7th day if weekly treatment is not completed. All participants will complete baseline assessments before treatment, six weekly treatments (except Group-3), a post-treatment assessment immediately and four-week after treatment. Randomly selected participants will complete an individual interview after treatment. Feedback will be gathered through a phone call to improve the intervention in the future.

DETAILED DESCRIPTION:
This study will be a pilot randomized control trial that examines the efficacy of guided and unguided transdiagnostic online self-help cognitive behavioral therapy for reducing symptoms of anxiety and depression in the Hong Kong adult resident population. Despite online self-help intervention has been widely recognized by its efficacy in improving depression and anxiety symptoms, the existing literature overlooks the mechanism of change and the potential predictors of online treatment outcome, as well as the effect of therapist's guidance on participants' treatment expectancy and its mediating effect on treatment outcome. However, the aforementioned research gaps are essential for optimizing the efficacy of online self-help interventions.

Prior to all study procedures, online informed consent with phone support will be obtained from potential participants. Around 96 eligible participants will be randomly assigned to either guided intervention group or unguided intervention group or waitlist control group in a ratio of 1:1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. No deception is necessary.

The participants in the guided intervention group will receive feedback calls (approximately 15 minutes) on participants' progress after each online self-help intervention session. The check-in includes treatment concepts clarification, homework checking, and technical issues solving. The check-ins will be delivered by a clinical psychology trainee or an undergraduate trained psychology student under the supervision of a clinical psychology professor. The participants in the unguided intervention group will not receive the aforementioned check-ins. The participants in both guided and unguided intervention groups will receive an email reminder and text message if the participants have not completed the required session of that week on the 5th, 6th, and 7th of the same week. Both technical supports are available for both groups. The waitlist unguided control group will not receive any online self-help intervention. All participants will complete a set of baseline assessments before the first session, a post-treatment assessment immediately after treatment, and a post-treatment assessment four-week after the treatment. Apart from the waitlist control group, both guided and unguided intervention groups will receive a total of six weekly online treatments. Randomly selected participants will complete an individual interview after treatment. Feedback will be gathered through a phone call or online feedback form to improve the intervention in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Have anxiety and/or depression symptoms, scoring 10 or above, in accordance with Patient Health Questionnaire (PHQ-9) or General Anxiety Disorder-7 (GAD-7);
2. Hong Kong residents aged 18-65;
3. Have access to the internet and have a valid email address for communication;
4. Able to read Chinese and type in Chinese or English; and
5. Willing to provide informed consent.

Exclusion Criteria:

1. Had received psychotherapy for depression and/or anxiety in the past 6 months;
2. Have reported the diagnosis of major psychiatric, bipolar disorder, medical or neurocognitive disorders, or have experienced dissociative symptoms that make participation infeasible or interfere with the adherence to the digital self-help intervention;
3. Will participate in another similar study/ other similar studies concurrently;
4. Any suicidal ideation (scoring above 2 in item 9 in PHQ-9)
5. Have reported substance abuse or dependence history;
6. Had changes in psychotropic drugs within 2 weeks before baseline assessment; and
7. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms - The Patient Health Questionnaire-9 (PHQ-9) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report measure that consists of 4-point Likert-scale questions that assess the severity of depressive symptoms. This measure reflects the DSM-IV diagnostic criteria of depression. Higher score means that the respondent has more depressive symptoms. Total score categories: 0-4 is no clinically significant depressive symptoms, 5-9 indicates mild depressive symptom,10-14 indicates moderate depressive symptoms, 15-19 indicates moderately severe depressive symptoms, 20-27 indicates extremely severe depressive symptom. This measure also shows good convergent validity with other measures and are widely used in mental health research (Beard et al., 2016; Kroenke et al., 2010)
Change in Anxiety Symptoms - The General Anxiety Disorder-7 (GAD-7) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The General Anxiety Disorder-7 (GAD-7) is a self-report measure to evaluate the severity of anxiety symptoms. This measure reflects the DSM-IV diagnostic criteria of anxiety. Total score categories: 0-4 is no clinically significant depressive symptoms, 5-9 indicates mild depressive symptom,10-14 indicates moderate depressive symptoms, 15-19 indicates moderately severe depressive symptoms, 20-27 indicates extremely severe depressive symptom. This measure also shows good convergent validity with other measures and are widely used in mental health research (Beard et al., 2016; Kroenke et al., 2010)

SECONDARY OUTCOMES:
Change in Quality-adjusted Life Years - The Short Form Six-Dimension (SF-6D) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The Short Form Six-Dimension (SF-6D) is a self-report measure that assesses health-related quality of life to estimate participant's quality-adjusted life years (QALYs). This instrument was validated in the Chinese population and widely applied in previous mental health research.
Change in Insomnia Severity Index (ISI) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  A 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem. Total score categories: 0-7 is no clinically significant insomnia, 8-14 is subthreshold insomnia,15-21 is clinical insomnia (moderate severity), and 22-28 is clinical insomnia (severe)
Change in the Perceived Stress Scale (PSS) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The PSS measures the perceived amount of stress experienced over the past month. The total score ranged from 0-40. Higher score means that the respondent has higher perceived stress level.
Change in emotional regulation strategies - Emotion Regulation Questionnaire (ERQ) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The Emotion Regulation Questionnaire (ERQ) is a self-report questionnaire that consists of 10 questions to assess how often the participants use cognitive reappraisal and expressive suppression as emotional regulation strategies. The total score ranged from 10-70. Higher score indicates that the respondent use cognitive reappraisal and expressive suppression as emotional regulation strategies more frequently.
Change in frequency of applying CBT-based skills - Frequency of Actions and Thoughts Scale (FATS) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  The Frequency of Actions and Thoughts Scale (FATS) is a self-report scale that assesses how frequent the participants apply the CBT-based skills they learned. The total score ranged from 0-48. Higher score means that the respondent has higher frequency of applying the CBT-based skills they learned.
Change in Positive Beliefs about Rumination Scale - Adapted Version (PBRS-A) | Baseline Assessment Phrase, Post-treatment Assessment Phrase (Immediately after Treatment), Post-treatment Assessment Phrase (Four-week after Treatment)
  Positive Beliefs about Rumination Scale (PBRS-A) is a 9-item instrument that measures positive belief on their rumination. The total score ranged from 9-36. Higher score means that the respondent has more positive beliefs about rumination.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong